CLINICAL TRIAL: NCT05087771
Title: In Hospital Administration of Extended-Release Naltrexone for Alcohol Use Disorder: A Pilot Study of Feasibility and Acceptability
Brief Title: In Hospital IM Naltrexone: A Pilot Study
Acronym: IM-NTX
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no longer randomized, drug being offered to all patients
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-4489
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Intervention Model Description: one group randomized to oral naltrexone; one group randomized to injectable naltrexone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral naltrexone (Active Comparator): patients will receive a 30 day supply of oral naltrexone 50 mg daily at hospital discharge. This medication was FDA approved in 1984 for the treatment of alcohol use disorder
  Interventions: Drug: oral naltrexone
- injectable naltrexone (Experimental): patient will receive 360 mg injection of naltrexone prior to hospital discharge
  Interventions: Drug: injectable naltrexone

INTERVENTIONS:
Drug: injectable naltrexone — 360 mg dose to be given prior to hospital discharge
  Other Names: Vivitrol
  Arms: injectable naltrexone
Drug: oral naltrexone — 50 mg tab dispense 30 day supply to be given at hospital discharge
  Arms: Oral naltrexone

SUMMARY:
This is a study in-hospital administration of injectable naltrexone vs. oral naltrexone. This is a pilot study to assess provider's and patient's acceptability to be randomized to oral vs. injectable naltrexone among hospitalized adults with alcohol use disorder.

DETAILED DESCRIPTION:
I. Hypotheses and Specific Aims: This proof of concept comparative effectiveness study seeks to pilot the administration of IM naltrexone among hospitalized adults with Diagnostic and Stastistical Manual-5 (DSM-5) diagnosis of alcohol use disorder at the University of Colorado Hospital and examine its acceptability and feasibility among patients and healthcare providers.

Study Aim 1: Test the feasibility and acceptability of recruiting, enrolling, and randomizing hospitalized patients, age 18 to 65 years old, with alcohol use disorder to treatment with in-hospital administration of IM naltrexone (n=30) versus oral naltrexone (n=60), both with linkage to outpatient follow-up.

Hypothesis 1: Outcomes such as recruitment rate, adverse events, and provider perception of the intervention's feasibility and acceptability in their clinical practice will help identify key lessons for a future comparative effectiveness study.

Study Aim 2: Estimate the combined 30-day readmission rate plus 30-day emergency department encounter rate for participants randomized to IM naltrexone vs. oral naltrexone.

Hypothesis 2: Combined 30-day readmission rate and emergency department encounter rate will be lower for IM naltrexone participants compared to oral naltrexone participants.

Study Aim 3: Estimate the 90-day treatment linkage rate for participants randomized to IM naltrexone vs. oral naltrexone.

Hypothesis 3: The 90-day treatment linkage rates will be higher for IM naltrexone participants compared to oral naltrexone participants.

Study Design and Research Methods Study Design: This study is pilot proof-of-concept, open-label comparative effectiveness trial of IM naltrexone vs. oral naltrexone among hospitalized adults with alcohol use disorder. Study outcomes include 1) an assessment of the feasibility to recruit, enroll, and randomize hospitalized patients to IM naltrexone (n=30) or oral naltrexone (n=60) and 2) an assessment of provider's perceived feasibility and acceptability to deliver the intervention. Comparative effectiveness outcomes include assessing the 1) combined 30-day readmission rate and 30-day emergency department encounter rate and 2) 90-day treatment linkage rates for participants randomized to IM naltrexone vs. oral naltrexone.

Study Site: The study will be conducted at the University of Colorado Hospital (UCH) where there is a weekday Addiction Consultation Service (ACS) who provides medication-assisted treatment for alcohol use disorder, including naltrexone, with facilitated linkage to post-discharge addiction care.

Recruitment: Eligible participants will be identified by an ACS team member through daily review of the ACS consultation list, focusing on consultation orders for "alcohol", e.g., alcohol withdrawal, and the sequela of alcohol use, trauma in the setting of alcohol intoxication, acute encephalopathy, and/or seizures, delirium tremens related to alcohol withdrawal. ACS attendings will complete routine addiction medicine care, including history taking, performing a physical exam, reviewing laboratory values, and a discussion of the assessment and plan, while considering the patient's alcohol use goals e.g., cut back, abstinence, no change in use, etc. If the patient meets criteria for an alcohol use disorder, the ACS attending will consider the use of naltrexone as medication-assisted treatment. If the patient expresses an interest in naltrexone, the attending will contact the one of the two addiction medicine team social workers or peer navigator, who is not involved in the patient's care, will approach the patient to inquire if the participants are interested in participating in the study. If the patient agrees, the participants will be consented and enrolled into the study and will be randomized to 2:1 to oral naltrexone or IM naltrexone. The ACS team member will alert the ACS attending who will either prescribe oral naltrexone to start during hospitalization with a 30-day prescription at discharge or who will administer IM naltrexone prior to hospital discharge. If the patient declines enrollment, the ACS attending will prescribe a 30-day supply of oral naltrexone. If a patient is interested in receiving IM naltrexone, the participants will be scheduled a follow-up appointment with a local clinic that provides this medication in the outpatient setting. All patients will be offered a follow-up appointment for ongoing treatment for their alcohol use disorder regardless of study enrollment.

Intervention: Participants will be randomized 2:1 to of oral naltrexone (n=60) oral naltrexone or IM naltrexone (n=30). Oral naltrexone is a once daily medication. IM naltrexone is dosed once monthly and is injected into the gluteal tissue. All participants will be scheduled a follow-up appointment with an addiction treatment provider or primary care provider between 30 to 90 days post hospital discharge, unless the participants decline the appointment.

The cost of oral naltrexone is covered by most insurance plans, including Colorado Medicaid, and is readily available in most pharmacies. For uninsured patients, the ACS team will work with the Atrium pharmacy and team social worker to obtain a voucher for medication coverage. This is the usual process for medication payment when a patient is unable to afford their medication co-pay or the cost of the medication at UCH. IM naltrexone is produced by Alkermes. Due to bundled insurance payments for hospitalizations, administration of IM naltrexone is prohibited for in-hospital administration at UCH (and at many hospitals) due to lack of reimbursement for services and product. In light of the potential treatment gap for hospitalized patients with alcohol use disorder, Alkermes created the "Hospital Inpatient Free Trail Program". This program allows for in-hospital administration of IM naltrexone which is provided free to the patient as a sample.

At the time of study enrollment, the ACS team member will ask a series of validated questions from the Addiction Severity Index Lite (ASI-Lite), a widely used instrument to assess the severity of problems related to substance use. The survey questions produce reliable and valid estimates of patient status in various life domains including 1) alcohol use, 2) medical health, 3) employment, and 4) illegal activity. These measure are mathematically derived and have shown reliability and validity in several settings. Composite scores will be assessed and reported for questions related to medical condition and alcohol use at baseline (see Appendix, Table 1 for ASI questions and composite questions). Assessments will be completed online using REDCap survey tools. Appendix, Table 1 lists baseline ASI-Lite questions to be asked.

Surveys to assess provider's perceived feasibility and acceptability of the intervention will be sent out prior to the study implementation, at study midpoint (when enrollment is 50% complete), and at study completion. The survey will be sent to all providers on the ACS (social workers, peer navigators, and physicians) (n=13). Surveys will be created and disseminated in REDCap and will be sent out in three waves to improve response rate. The survey will include sections where ACS team members can type in their thoughts and perceptions of the intervention and make any recommendations for improvement. These data will be qualitative, in contrast to the quantitative survey data, and will be used to inform our future comparative effectiveness trial.

Data Collection Tools: REDCap or the Electronic Helath Record (EHR) via Health Data Compass.

Data Analysis Plan:

Baseline Comparison of Treatment Groups: Participant's characteristics and baseline clinical data will be tabulated, and differences between IM vs. oral naltrexone groups will be assessed using a Fisher's Exact Test for categorical variables and Wilcoxon rank-sum tests and Chi-squared tests for continuous variables.

Propensity Score Inverse Probability of Treatment Weighting: The investigators will use inverse probability of treatment weighting (IPTW) based on the propensity score to reduce bias by ensuring that participants who are randomized to IM naltrexone (n=30) vs. oral naltrexone (n=60) will have comparable covariate distributions. Propensity scores will be calculated from a multivariable logistic regression model with a binary outcome of IM naltrexone treatment or oral naltrexone treatment. Variables shown in Appendix, Table 1 will be included if the variables are significantly associated with both IM naloxone treatment and the outcome or with the outcome only. Significance will be assessed based on clinical judgement and bivariate statistical analysis (p-value < 0.05). If highly collinear variables are included in the model, variables associated with both IM naloxone treatment and the outcome will be preferred over those only associated with the outcome. Weights will be stabilized to more accurately estimate variance if a small number of weights become especially large and influential due to particularly low or high propensity scores. After applying weights, covariate distributions will be compared between the group receiving IM naltrexone and the group receiving oral naltrexone to ensure that confounding variable distributions are approximately balanced between groups.

Once IM naltrexone and oral naltrexone groups are matched, the investigators will assess comparative effectiveness outcomes, 30-day all cause hospitalization rates+ 30-day emergency department encounter rates by IM vs. oral naltrexone, and 90-day post discharge linkage rates by IM vs. oral naltrexone group. This pilot study is not sufficiently powered for hypothesis testing on these outcomes. By way of example, the use of 30 participants compared to 60 participant controls yields just 40% power to detect a 50% relative difference in readmission using a pilot appropriate alpha of 10%.36 Regardless, the readmission risk differences will be evaluated using multiple logistic regression to assess the association of treatment on 30-day combined readmissions and emergency department encounter rates. The investigators will use multiple logistic regression to assess the association between IM naltrexone or oral naltrexone on 90-day addiction treatment linkage. These findings will provide parameter estimates that can inform a future sample size calculation in a larger effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

Participants will include hospitalized adults, aged 18 to 65 years old, who receive care from the ACS during their hospitalization and who meet DSM - 5 criteria for alcohol use disorder.

Exclusion Criteria:

Naltrexone is contraindicated in acute hepatitis or liver failure and its use in patients with active liver disease must be carefully considered in light of the potential for hepatotoxic effects.23 It is also contraindicated in patients taking opioids for pain due to its antagonism at the opioid receptor.23 The investigators will exclude people who meet the following criteria:

* Liver function test (AST/ALT) more than five times the upper limit of normal
* Decompensated liver failure defined as use of lactulose for prevention of hepatic encephalopathy, ascites, use of spironolactone and/or lasix for ascites, presence of hepatic encephalopathy, International Normalized Ratio (INR) >2, or thrombocytopenia in the setting of known liver disease
* Renal failure, defined as a glomerular filtration rate of <30 ml/min
* On opioids for acute or chronic pain at time of study enrollment
* Pregnancy, IM naltrexone is not FDA approved in pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months
  The investigators will assess recruitment rate for IM naltrexone and oral naltrexone
  o Recruitment is defined as ([number of participants enrolled / number of participants enrolled approached] / 12 months)

SECONDARY OUTCOMES:
II. Acceptability and Feasibility Measures | prior to study implementation and after 50% enrollment is completed, approximately 6 months from study start date
  The investigators will use survey questions to assess acceptability and feasibility with responses measured using a 5-point Likert scale titled "Intervention Acceptability and Feasibility". The scale ranges include: (1) completely disagree [minimum value], (2) disagree, (3) neither agree nor disagree, (4) agree, (5) completely agrees [maximum value]). Maximum value (5) means the intervention is the most acceptable and the most feasible.
III. Comparative Effectiveness: Combined all-cause 30-day readmission rate + all cause 30-day emergency department encounter rate. | 30 days from time of last person enrolled in study
  Combined all-cause 30-day readmission rate + all cause 30-day emergency department encounter rate Data assessing measures III and IV will be obtained from Health Data Compass at University of Colorado27 which includes data obtained from the All Payer Claims Dataset (APCD)28 and University of Colorado health related-encounters.
IV. Comparative Effectiveness: 90-day addiction treatment encounter rate for participants randomized to IM vs. oral naltrexone | 90 days from time of last person enrolled in study
  90-day addiction treatment encounter rate for participants randomized to IM vs. oral naltrexone defined as "documentation of ≥ 1 healthcare encounters with an associated International Statistical Classification of Diseases and Related Health Problems (ICD)-code for alcohol use disorder (F10.X) identified within 90 days following the index hospitalization"
  o Data assessing measures III and IV will be obtained from Health Data Compass at University of Colorado27 which includes data obtained from the All Payer Claims Dataset (APCD)28 and UCHealth related-encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lynn Calcaterra, MD, MPH, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
This is not part of our study protocol and will not be included as part of the consent for study participation.

REFERENCES:
- [Result] Health UDo, Services H, Control CfD, Prevention, Statistics NCfH. Bridged-race population estimates, United States July 1st resident population by state, county, age, sex, bridged-race, and Hispanic origin. Compiled from. 1990;1999:2000-2009.
- [Result] Abuse S. Mental Health Services Administration.(2017). Key substance use and mental health indicators in the United States: Results from the 2016 National Survey on Drug Use and Health (HHS Publication No. SMA 17-5044, NSDUH Series H-52). Rockville, MD: Center for Behavioral Health Statistics and Quality. Substance Abuse and Mental Health Services Administration Retrieved from https://www samhsa gov/data. 2018.
- [Result] Laramee P, Leonard S, Buchanan-Hughes A, Warnakula S, Daeppen JB, Rehm J. Risk of All-Cause Mortality in Alcohol-Dependent Individuals: A Systematic Literature Review and Meta-Analysis. EBioMedicine. 2015 Sep 2;2(10):1394-404. doi: 10.1016/j.ebiom.2015.08.040. eCollection 2015 Oct. PMID 26629534
- [Result] Roerecke M, Rehm J. Alcohol use disorders and mortality: a systematic review and meta-analysis. Addiction. 2013 Sep;108(9):1562-78. doi: 10.1111/add.12231. Epub 2013 May 29. PMID 23627868
- [Result] Chen C, Yoon Y. Trends in Alcohol-Related Morbidity Among Community Hospital Discharges, United States, 2000-2015. Surveillance Report# 112. Arlington, VA. 2018.
- [Result] Jonas DE, Amick HR, Feltner C, Bobashev G, Thomas K, Wines R, Kim MM, Shanahan E, Gass CE, Rowe CJ, Garbutt JC. Pharmacotherapy for adults with alcohol use disorders in outpatient settings: a systematic review and meta-analysis. JAMA. 2014 May 14;311(18):1889-900. doi: 10.1001/jama.2014.3628. PMID 24825644
- [Result] Kirchoff RW, Mohammed NM, McHugh J, Markota M, Kingsley T, Leung J, Burton MC, Chaudhary R. Naltrexone Initiation in the Inpatient Setting for Alcohol Use Disorder: A Systematic Review of Clinical Outcomes. Mayo Clin Proc Innov Qual Outcomes. 2021 Apr 8;5(2):495-501. doi: 10.1016/j.mayocpiqo.2021.01.013. eCollection 2021 Apr. PMID 33997645
- [Result] Jaffe AJ, Rounsaville B, Chang G, Schottenfeld RS, Meyer RE, O'Malley SS. Naltrexone, relapse prevention, and supportive therapy with alcoholics: an analysis of patient treatment matching. J Consult Clin Psychol. 1996 Oct;64(5):1044-53. doi: 10.1037//0022-006x.64.5.1044. PMID 8916634
- [Result] O'Malley SS, Jaffe AJ, Chang G, Schottenfeld RS, Meyer RE, Rounsaville B. Naltrexone and coping skills therapy for alcohol dependence. A controlled study. Arch Gen Psychiatry. 1992 Nov;49(11):881-7. doi: 10.1001/archpsyc.1992.01820110045007. PMID 1444726
- [Result] Volpicelli JR, Alterman AI, Hayashida M, O'Brien CP. Naltrexone in the treatment of alcohol dependence. Arch Gen Psychiatry. 1992 Nov;49(11):876-80. doi: 10.1001/archpsyc.1992.01820110040006. PMID 1345133
- [Result] Anton RF, Moak DH, Waid LR, Latham PK, Malcolm RJ, Dias JK. Naltrexone and cognitive behavioral therapy for the treatment of outpatient alcoholics: results of a placebo-controlled trial. Am J Psychiatry. 1999 Nov;156(11):1758-64. doi: 10.1176/ajp.156.11.1758. PMID 10553740
- [Result] Monti PM, Rohsenow DJ, Swift RM, Gulliver SB, Colby SM, Mueller TI, Brown RA, Gordon A, Abrams DB, Niaura RS, Asher MK. Naltrexone and cue exposure with coping and communication skills training for alcoholics: treatment process and 1-year outcomes. Alcohol Clin Exp Res. 2001 Nov;25(11):1634-47. PMID 11707638
- [Result] Croop RS, Faulkner EB, Labriola DF. The safety profile of naltrexone in the treatment of alcoholism. Results from a multicenter usage study. The Naltrexone Usage Study Group. Arch Gen Psychiatry. 1997 Dec;54(12):1130-5. doi: 10.1001/archpsyc.1997.01830240090013. PMID 9400350
- [Result] Fairbanks J, Umbreit A, Kolla BP, Karpyak VM, Schneekloth TD, Loukianova LL, Sinha S. Evidence-Based Pharmacotherapies for Alcohol Use Disorder: Clinical Pearls. Mayo Clin Proc. 2020 Sep;95(9):1964-1977. doi: 10.1016/j.mayocp.2020.01.030. Epub 2020 May 20. PMID 32446635
- [Result] Garbutt JC, Kranzler HR, O'Malley SS, Gastfriend DR, Pettinati HM, Silverman BL, Loewy JW, Ehrich EW; Vivitrex Study Group. Efficacy and tolerability of long-acting injectable naltrexone for alcohol dependence: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1617-25. doi: 10.1001/jama.293.13.1617. PMID 15811981
- [Result] Johnson BA. Naltrexone long-acting formulation in the treatment of alcohol dependence. Ther Clin Risk Manag. 2007 Oct;3(5):741-9. PMID 18472999
- [Result] Murphy CE 4th, Wang RC, Montoy JC, Whittaker E, Raven M. Effect of extended-release naltrexone on alcohol consumption: a systematic review and meta-analysis. Addiction. 2022 Feb;117(2):271-281. doi: 10.1111/add.15572. Epub 2021 Jun 28. PMID 34033183
- [Result] Wei J, Defries T, Lozada M, Young N, Huen W, Tulsky J. An inpatient treatment and discharge planning protocol for alcohol dependence: efficacy in reducing 30-day readmissions and emergency department visits. J Gen Intern Med. 2015 Mar;30(3):365-70. doi: 10.1007/s11606-014-2968-9. Epub 2014 Aug 5. PMID 25092008
- [Result] Financing CDoHCPa. Colorado Hospital Transformation Program. Colorado Office State Web Portal. https://hcpf.colorado.gov/colorado-hospital-transformation-program. Published 2021. Accessed September 16, 2021
- [Result] Calcaterra SL, McBeth L, Keniston AM, Burden M. The Development and Implementation of a Hospitalist-Directed Addiction Medicine Consultation Service to Address a Treatment Gap. J Gen Intern Med. 2022 Apr;37(5):1065-1072. doi: 10.1007/s11606-021-06849-8. Epub 2021 May 19. PMID 34013473
- [Result] Grant BF, Goldstein RB, Saha TD, Chou SP, Jung J, Zhang H, Pickering RP, Ruan WJ, Smith SM, Huang B, Hasin DS. Epidemiology of DSM-5 Alcohol Use Disorder: Results From the National Epidemiologic Survey on Alcohol and Related Conditions III. JAMA Psychiatry. 2015 Aug;72(8):757-66. doi: 10.1001/jamapsychiatry.2015.0584. PMID 26039070
- [Result] Administration SAaMHS. Incorporating Alcohol Pharmacotherapies into Medical Practice: Treatment Improvement Protcol (TIP) Series, No. 49. Rockville, MD2009.
- [Result] Alkermes. Alkermes Hospital Inpatient Free Trail Program. Alkermes. https://www.alkermeshospitalprogram.com/. Published 2021. Accessed September 16, 2021.
- [Result] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Result] Weiner BJ, Lewis, C. C., Stanick, C., Powell, B. J., Dorsey, C. N., Clary, A. S., Boynton, M. H., & Halko, H. Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), & Feasibility of Intervention Measure. Frank Porter Graham Child Development Institute;2017.
- [Result] Compass HD. Health Data Compass. https://pub.healthdatacompass.org/data-delivery-services/health-data-compass-resources. Published 2019. Accessed September 14, 2021
- [Result] (CIVHC) CfIViH. CO APCD Overview. https://www.civhc.org/get-data/co-apcd-info/. Published 2021. Accessed September 14, 2021.
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Cacciola JS, Alterman AI, McLellan AT, Lin YT, Lynch KG. Initial evidence for the reliability and validity of a "Lite" version of the Addiction Severity Index. Drug Alcohol Depend. 2007 Mar 16;87(2-3):297-302. doi: 10.1016/j.drugalcdep.2006.09.002. Epub 2006 Oct 11. PMID 17045423
- [Result] McLellan A, Cacciola J, Zanis D. The addiction severity index-lite. Center for the Studies on Addiction, University of Pennsylvania/Philadelphia VA Medical Center. 1997.
- [Result] McLellan AT, Kushner H, Metzger D, Peters R, Smith I, Grissom G, Pettinati H, Argeriou M. The Fifth Edition of the Addiction Severity Index. J Subst Abuse Treat. 1992;9(3):199-213. doi: 10.1016/0740-5472(92)90062-s. PMID 1334156
- [Result] McGahan PL, Griffith JA, Parente R, McLellann AT. Composite scores manual. Treatment Research Institute Philadelphia, PA. 1986.
- [Result] Brookhart MA, Schneeweiss S, Rothman KJ, Glynn RJ, Avorn J, Sturmer T. Variable selection for propensity score models. Am J Epidemiol. 2006 Jun 15;163(12):1149-56. doi: 10.1093/aje/kwj149. Epub 2006 Apr 19. PMID 16624967
- [Result] Cervantes L, Tuot D, Raghavan R, Linas S, Zoucha J, Sweeney L, Vangala C, Hull M, Camacho M, Keniston A, McCulloch CE, Grubbs V, Kendrick J, Powe NR. Association of Emergency-Only vs Standard Hemodialysis With Mortality and Health Care Use Among Undocumented Immigrants With End-stage Renal Disease. JAMA Intern Med. 2018 Feb 1;178(2):188-195. doi: 10.1001/jamainternmed.2017.7039. PMID 29255898
- [Result] Lee EC, Whitehead AL, Jacques RM, Julious SA. The statistical interpretation of pilot trials: should significance thresholds be reconsidered? BMC Med Res Methodol. 2014 Mar 20;14:41. doi: 10.1186/1471-2288-14-41. PMID 24650044